CLINICAL TRIAL: NCT01305811
Title: Acupuncture in the Treatment of Gulf War Illness
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New England School of Acupuncture (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lisa Conboy, Director of Research, New England School of Acupuncture
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GW080059(W81XWH-09-2-0064)
Record Dates: First submitted 2011-02-24; First posted 2011-03-01 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-05

CONDITIONS: Persian Gulf Syndrome
Keywords: Complex Medical Illness; Gulf War Illness; Veteran
MeSH Terms: conditions — Persian Gulf Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bi-weekly acupuncture treatment (Experimental): Bi-weekly acupuncture treatment
  Interventions: Device: Acupuncture
- Wait list (Active Comparator): Wait list for 2 months followed by weekly acupuncture for 4 months
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — Sterile insertive needles are applied by licensed, experienced practitioners.

SUMMARY:
This unblinded Phase II clinical trial tested the effects of individualized acupuncture treatments offered in extant acupuncture practices in the community; practitioners had at least 5 years of experience plus additional training provided by the study. Veterans with diagnosed symptoms of Gulf War Illness were randomized to either six months of biweekly acupuncture treatments (group 1, n=52) or 2 months of waitlist followed by weekly acupuncture treatments (group 2, n=52). Measurements were taken at baseline, 2, 4 and 6 months. The primary outcome is the SF-36 physical component scale score (SF-36P).

DETAILED DESCRIPTION:
Gulf War Illness (GWI) is a complex, poorly understood illness characterized by many symptoms, including fatigue after exertion, sleep and mood problems, difficulty concentrating, difficulty thinking and finding words, and musculoskeletal pain. Individuals often present with many symptoms, some of them severe and disabling, and with additional medical diagnoses, including chronic fatigue syndrome, fibromyalgia, irritable bowel syndrome, digestive complaints, and mood-related psychiatric disorders, such as depression, posttraumatic stress disorder, and other anxiety disorders. More than 100,000 veterans of the first Gulf War (Operation Desert Shield/Storm, 1990-1991) out of 700,000 US service personnel deployed to the Persian Gulf have presented with medical complaints through programs established to address the problem, which came to be called chronic multisymptom illness (CMI). Groups of veterans in the United Kingdom, Canada, and Australia have been identified with similar problems. The veterans have received treatment directed at their symptoms, but at 5- and 10-year follow-ups, many reported their symptoms remained, some of them severe and disabling. Clearly, an effective treatment for these conditions would be of great benefit to those who were injured during their military service.

The cause of CMI is unknown, and the symptoms can not be explained by physical and laboratory examinations. Several factors have been considered, including exposure to vaccines, chemicals likely to be encountered in combat (chemical weapons, smoke, pesticides) and stress related to military service, deployment, and combat. After investigation by the Centers for Disease Control (CDC), researchers suspect that the symptoms reflect a range of injuries to the nervous system. It may be that the factors that led to these injuries were not specific to the Persian Gulf region, and that veterans of the current war in Iraq and Afghanistan, as well as active duty personnel, are exposed to similar stressors and will benefit from an investigation of CMI and its treatment.

The goal of this study is to help identify whether acupuncture is an effective treatment for Gulf War Syndrome. Acupuncture is likely to be helpful in treating GWI because it has already been used successfully to reduce many of its key symptoms - fatigue, irritability, anxiety, insomnia, and pain. Acupuncture treatment is designed to treat each individual's symptoms making it very well suited for treating the varied symptoms of GWI. Veterans will receive care that is directed specifically at their most distressing symptom. Although the specific etiology of CMI is unknown, acupuncture's analgesic and anti-inflammatory effects are likely to be helpful. Acupuncture seems to work, in part, on peripheral nerves near the site of injury, in the brain, central nervous system, and on the endocrine system, in ways that promote the body's own efforts to reduce pain and heal even chronic injuries. Numerous studies have shown acupuncture is well tolerated by patients, safe, and cost-effective compared to routine care. Acupuncture will be provided by licensed acupuncturists with at least 5 years of clinical experience, who have received 20-hours of training related to symptoms of GWI.

Subjects were recruited via local advertisements and direct mailing to veterans on the Defense Manpower Data Center (http://www.virec.research.va.gov/Non-VADataSources/DMDC.htm). Through questionnaires, physician assessment, and medical histories, the investigators measured the severity of symptoms before beginning treatment, and after 2, 4 and 6 months of treatment. One group of patients received acupuncture evaluation and treatment twice per week for 6 months. A second group, for comparison purposes, will be monitored on a wait list for 2 months, and will then be offered weekly acupuncture for 4 months. Based on previous acupuncture research on fatigue, stress, and pain, the investigators expect this length of treatment will be enough for patients to receive significant benefit. The investigators also planed to collect samples of blood from our volunteers that will help identify possible disease mechanisms for the illness and track the effects of treatment.

ELIGIBILITY:
Inclusion

1. deployed to the "Gulf Theater of operations, as defined by 38 CFR 3.317, includes Iraq, Kuwait, Saudi Arabia, Bahrain, Qatar, the United Arab Emirates, Oman, the Gulf of Aden, the Gulf of Oman, the Persian Gulf, the Arabian Sea, the Red Sea, and the airspace above all of these locations" between August 1990 and the present date,
2. they have at least 2 of the following symptoms from the 3 CDC clusters of symptom that have lasted for more than 6 months. Each symptom cluster must be characterized as "mild-moderate" or "severe" with at least one symptom in each cluster required to be severe. The clusters are:

A-Fatigability

* fatigue 24 hours or more after exertion B-Mood and Cognition
* feeling depressed or
* feeling irritable or
* difficulty thinking or concentrating or
* feeling worried, tense, anxious or
* problems finding words or
* problems getting to sleep C-Musculoskeletal
* joint pain or muscle pain

Exclusion:

* Currently enrolled in another clinical trial
* Have another disease that likely could account for the symptoms, as determined by our Medical Monitor
* Severe psychiatric illness (in the last 2 years psychiatric hospitalization, suicidal attempt, alcohol or substance abuse, use of antipsychotic medication) as measured by the Primary Care Evaluation of Mental Disorder (Prime MD).
* Unable to complete the protocol on based on the evaluation of the Medical Monitor

Min Age: 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Conboy, ScD, Principal Investigator — New England School of Acupuncture
Locations (1):
- New England School of Acupuncture, Newton, Massachusetts, United States

REFERENCES:
- [Derived] Conboy L, Gerke T, Hsu KY, St John M, Goldstein M, Schnyer R. The Effectiveness of Individualized Acupuncture Protocols in the Treatment of Gulf War Illness: A Pragmatic Randomized Clinical Trial. PLoS One. 2016 Mar 31;11(3):e0149161. doi: 10.1371/journal.pone.0149161. eCollection 2016. PMID 27031099

RESULTS

PARTICIPANT FLOW:
Groups:
- Bi-weekly Acupuncture Treatment: Veterans with diagnosed symptoms of Gulf War Illness were randomized to six months of biweekly acupuncture treatments.
- Wait List: Veterans with diagnosed symptoms of Gulf War Illness were randomized to 2 months of waitlist followed by weekly acupuncture treatments for 4 months.
Period: Overall Study
Arm/Group | Bi-weekly Acupuncture Treatment | Wait List
Started | 52 | 52
Completed | 44 | 41
Not Completed | 8 | 11

BASELINE CHARACTERISTICS:
Groups:
- Bi-weekly Acupuncture Treatment: Bi-weekly acupuncture treatment for 6 months
- Wait List: Wait list for 2 months then weekly acupuncture for four months
- Total: Total of all reporting groups
Arm/Group | Bi-weekly Acupuncture Treatment | Wait List | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 52 | 104
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (9.9) | 48.2 (3.5) | 48.2 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 45 | 45 | 90
Region of Enrollment [Number; unit: participants]
  United States | 52 | 52 | 104

OUTCOME MEASURES:

1. Primary Outcome: SF-36P
Description: Ten items addressing physical functioning which are part of a short-form health survey with 36 questions. Scores range between 0 and 100 with higher scores indicating better function.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Bi-Weekly Acupuncture; Wait List Then Weekly Acupuncture: group mean SF-36 P score at 6 months
Arm/Group | Bi-Weekly Acupuncture | Wait List Then Weekly Acupuncture
Number analyzed (Participants) | 44 | 41
units on a scale | 73.7 [67.7 to 79.8] | 64.3 [57.1 to 71.4]
Statistical Analysis 1: Comparison: Bi-Weekly Acupuncture vs Wait List Then Weekly Acupuncture; Test type: Superiority or Other; p = 0.03, general estimating equations

2. Other Pre Specified Outcome: SF-36P
Description: as for outcome 1
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Wait List: Wait list for 2 months.
  Acupuncture: Sterile insertive needles are applied by licensed, experienced practitioners.
Arm/Group | Bi-weekly Acupuncture Treatment | Wait List
Number analyzed (Participants) | 50 | 50
units on a scale | 0.32 (16.8) | 4.53 (14.8)
Statistical Analysis 1: Comparison: Bi-weekly Acupuncture Treatment vs Wait List; In our original proposal to the funder, to protect our main outcome from possibly large attrition, we proposed to initially test mean differences between groups following 2 months of treatment or wait list using Student's t-tests at an alpha=0.05; Test type: Superiority or Other; p = 0.22, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 years 5 months
Description: All potential adverse events which occurred in either study arm were reviewed by the study's medical monitor. Serious and/or unexpected events were reported to the Main IRB and the funder's review office (Army Human Research Protection Office (HRPO)).
Groups:
- Bi-Weekly Acupuncture: Bi-Weekly Acupuncture for 6 months
  1 serious unexpected adverse event in the biweekly group: Subject's practitioner was told by subject of a suicide attempt. Case was reviewed and the medical monitor and identified as needing follow up. Subject was hospitalized for observation, released to his daughter's custody. Both the VA and the Crisis Center were in touch with him on Feb 27th and are making arrangements to take him, (patient reported), either in patient or into a program. He had a follow-up appointment Feb 28th at the VA and he was hospitalized at this time and is currently hospitalized.
  The practitioner will also follow up with subject's PCP.
- Wait List: Wait list for 2 months followed by 4 months of weekly acupuncture
  No Adverse events were reported in the Wait list group
Arm/Group | Bi-Weekly Acupuncture | Wait List
Serious Adverse Events (participants affected / at risk) | 1/52 | 0/52
Other Adverse Events (participants affected / at risk) | 1/52 | 0/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bi-Weekly Acupuncture (N=52) | Wait List (N=52)
Serious unexpected (Social circumstances) | 1 | 0 — Subject's practitioner was told by subject of a suicide attempt.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bi-Weekly Acupuncture (N=52) | Wait List (N=52)
Pain on needling (Social circumstances) | 1 (52) | 0 — Subject is experiencing pain at one of the acupuncture points that was needled and this pain has lasted longer than is typical.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No